CLINICAL TRIAL: NCT01956240
Title: Phase 4 Effects of a Stretching Protocol for the Pectoralis Minor Muscle on This Resting Length and on the 3D Kinematics of the Scapula During Arm Flexion in Asymptomatic Subjects and Patients With Impingement Syndrome
Brief Title: Effects of a Pectoralis Minor Muscle Stretching Protocol
Acronym: PMISP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universidade Federal de Sao Carlos (Other)
Collaborators: Universidade Metodista de Piracicaba (Other)
Responsible Party: Principal Investigator, Dayana Patricia Rosa, Universidade Federal de São Carlos, Universidade Federal de Sao Carlos
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 100/12
Record Dates: First submitted 2013-09-21; First posted 2013-10-08 (Estimated); Results first posted 2015-02-12 (Estimated); Last update posted 2015-05-19 (Estimated); Status verified 2015-05

CONDITIONS: Shoulder Pain
Keywords: shoulder; pectoralis minor; stretching; scapular kinematics
MeSH Terms: conditions — Shoulder Pain

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Stretching-Asymptomatic subjects (Experimental): The stretching will be performed with the subject standing, with 90° of arm abduction and 90° of elbow flexion and palm on a flat planar surface. The subject then will place the leg opposite to the flat surface in front of the other with slight knee flexion and tilt the trunk forward like a rigid block and rotate it slightly increasing the horizontal abduction at the shoulder. This procedure will be done 4 times for 1 min and 30s interval between repetitions.
  Interventions: Procedure: Stretching-Asymptomatic subjects
- Stretching-Subjects with shoulder pain (Experimental): The stretching will be performed with the subject standing, with 90° of arm abduction and 90° of elbow flexion and palm on a flat planar surface. The subject then will place the leg opposite to the flat surface in front of the other with slight knee flexion and tilt the trunk forward like a rigid block and rotate it slightly increasing the horizontal abduction at the shoulder. This procedure will be done 4 times for 1 min and 30s interval between repetitions.
  Interventions: Procedure: Stretching-Subjects with shoulder pain

INTERVENTIONS:
Procedure: Stretching-Asymptomatic subjects — The stretching will be performed with the subject standing, with 90° of arm abduction and 90° of elbow flexion and palm on a flat planar surface. The subject then will place the leg opposite to the flat surface in front of the other with slight knee flexion and tilt the trunk forward like a rigid block and rotate it slightly increasing the horizontal abduction at the shoulder. This procedure will be done 4 times for 1 min and 30s interval between repetitions.
  Arms: Stretching-Asymptomatic subjects
Procedure: Stretching-Subjects with shoulder pain — The stretching will be performed with the subject standing, with 90° of arm abduction and 90° of elbow flexion and palm on a flat planar surface. The subject then will place the leg opposite to the flat surface in front of the other with slight knee flexion and tilt the trunk forward like a rigid block and rotate it slightly increasing the horizontal abduction at the shoulder. This procedure will be done 4 times for 1 min and 30s interval between repetitions.
  Arms: Stretching-Subjects with shoulder pain

SUMMARY:
The purpose of this study is to verify the effects of a stretching protocol for the pectoralis minor muscle on its resting length and on the 3D kinematics of the scapula during arm flexion in asymptomatic subjects and patients with impingement syndrome with shortened pectoralis minor.

DETAILED DESCRIPTION:
Fifty subjects (25 symptomatic and 25 asymptomatic for shoulder pain) will be recruited. All of them will be initially assessed twice with one week between the assessments. On each day, they will complete two questionnaires (DASH and SPADI) to assess pain and shoulder function. The resting length of the pectoralis minor muscle and scapular kinematics data during arm flexion will also be measured using an electromagnetic tracking system. Initially, the resting length of the pectoralis minor will be measured, and then 3 repetitions of arm elevation in the sagittal plane will be completed. The stretching protocol will be performed daily for 6 weeks. The stretching will be performed with the subject standing, with 90° of arm abduction and 90° of elbow flexion and palm on a flat planar surface. The subject then will place the leg opposite to the flat surface in front of the other with slight knee flexion and tilt the trunk forward like a rigid block and rotate it slightly increasing the horizontal abduction at the shoulder. This procedure will be done 4 times for 1 min and 30s interval between repetitions. After the 6 weeks, the subject will have the same variables from the initial assessments reassessed. For the questionnaires and length of pectoralis minor a two-way ANOVA for repeated measures will be used to check the main effects of group and evaluation and whether there is interaction between them. For scapular internal/external rotation, upward/downward rotation, and tilt anterior/posterior a three-way ANOVA for repeated measures will use to analyze the main effects of group (symptomatic and asymptomatic), elevation angle of the arm (30°, 60°, 90° and 120°) and evaluation (1, 2 and 3) and whether there is evaluation x group x angle interaction. A p value less than 0.05 will be considered significant.

ELIGIBILITY:
Inclusion Criteria:

Asymptomatic subjects were included if they did not have any positive test for SIS.

The subjects with shoulder pain were included if:

1. they had history of shoulder, at least one week;
2. 18 - 45 years;
3. range of motion > 150° evaluated with digital inclinometer;
4. one or more impingement tests positive - Neer (Neer, 1972), Hawkins (Hawkins and Kennedy, 1980) and Jobe (Jobe and Moynes, 1982) - associated with painful arc during arm elevation, or during external rotation with 90° of arm elevation;
5. Individuals from both groups also had to present with shortened PM muscle length.

Exclusion Criteria:

Individuals from both groups were excluded if they:

1. BMI (body mass index) > 28kg/m2;
2. irradiated shoulder pain;
3. scoliosis;
4. history of shoulder pain with beginning traumatic;
5. history of fracture or surgery in upper limb and rotator cuff;
6. systemic illnesses;
7. tape allergy;
8. were pregnant;
9. physiotherapy at least 6 months.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 97 (Actual)
Dates: Start 2013-06; Primary Completion 2013-08 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dayana Rosa, PT, Principal Investigator — UNIMEP
Locations (1):
- UFSCar, São Carlos, São Paulo, Brazil

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Fliers posted in the local university setting and community were used to recruit symptomatic individuals, between february of 2012 and January of 2014. Asymptomatic individuals were recruited through personal contacts of the investigators.
Pre-assignment Details: If participants did not come back to second evaluation, they were not assignments to groups.
Groups:
- Asymptomatic Subjects; Subjects With Shoulder Pain: The stretching will be performed with the subject standing, with 90° of arm abduction and 90° of elbow flexion and palm on a flat planar surface. The subject then will place the leg opposite to the flat surface in front of the other with slight knee flexion and tilt the trunk forward like a rigid block and rotate it slightly increasing the horizontal abduction at the shoulder. This procedure will be done 4 times for 1 min and 30s interval between repetitions.
Period: Overall Study
Arm/Group | Asymptomatic Subjects | Subjects With Shoulder Pain
Started | 48 | 49
Completed | 25 | 25
Not Completed | 23 | 24
Not completed — Lost to Follow-up | 6 | 20
Not completed — Adverse Event | 17 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Asymptomatic Subjects | Subjects With Shoulder Pain | Total
Number analyzed (Participants) | 48 | 49 | 97
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 48 | 49 | 97
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 28 | 54
  Male | 22 | 21 | 43
Region of Enrollment [Number; unit: participants]
  Brazil | 48 | 49 | 97

OUTCOME MEASURES:

1. Primary Outcome: Pectoralis Minor Length After Pectoralis Minor Stretching Protocol
Description: The change of the pectoralis minor muscle will be evaluated with a tape measure and electromagnetic device. The length of the muscle will be recorded in centimeters.
Time Frame: 6 weeks after stretching
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | Asymptomatic Subjects | Subjects With Shoulder Pain
Number analyzed (Participants) | 48 | 49
centimeters | 16.38 (1.46) | 16.87 (1.90)
Statistical Analysis 1: Comparison: Asymptomatic Subjects vs Subjects With Shoulder Pain; Test type: Superiority or Other; p < 0.05, ANOVA; A 1-way repeated measures ANOVA was used to assess for possible differences among evaluations in each group separately for pectoralis minor length; Median Difference (Final Values) = 0.51, Standard Deviation 1.90

2. Secondary Outcome: Scapular Kinematics After Pectoralis Minor Stretching Protocol
Description: The scapular kinematics will be evaluated with electromagnetic device. The changes in the scapular kinematics will be described in degrees.
Time Frame: 6 weeks of stretching
Measure: Mean (Standard Deviation); unit: degree
Arm/Group | Asymptomatic Subjects | Subjects With Shoulder Pain
Number analyzed (Participants) | 25 | 25
degree | 30 (5) | 40 (5)
Statistical Analysis 1: Comparison: Asymptomatic Subjects vs Subjects With Shoulder Pain; Test type: Superiority or Other; p > 0.05, ANOVA; Separate 2-way repeated measures ANOVAs were used to test for interactions of angle x evaluation (1,2,3) and for main effects of evaluation; Median Difference (Final Values) = 5

ADVERSE EVENTS:
Arm/Group | Asymptomatic Subjects | Subjects With Shoulder Pain
Serious Adverse Events (participants affected / at risk) | 23/48 | 24/49
Other Adverse Events (participants affected / at risk) | 15/48 | 7/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Asymptomatic Subjects (N=48) | Subjects With Shoulder Pain (N=49)
Desistance (Social circumstances) | 23 | 24 — Forty seven participants left this study because personal reasons.
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Asymptomatic Subjects (N=48) | Subjects With Shoulder Pain (N=49)
No shortened pectoralis minor (Musculoskeletal and connective tissue disorders) | 15 | 7 — Fifteen participants did not present shortening of pectoralis minor.

LIMITATIONS AND CAVEATS:
1. Participants may not have maximally elongated muscle;
2. Linear measurements such as that used to quantify muscle length cannot represent real structural changes;
3. Only chronic pain was evaluated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No